CLINICAL TRIAL: NCT01465373
Title: Comparison of the Effectiveness of Micronized Vaginal Progesterone (Endometrin, Ferring) Vs. Progesterone in Oil for Luteal Phase Support in Donor Egg Recipient IVF Cycles Utilizing Previously Vitrified Donor Oocytes
Brief Title: Vaginal Progesterone Versus Progesterone in Oil in Donor Egg Recipient In Vitro Fertilization Cycles Utilizing Vitrified Donor Eggs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fertility Centers of Illinois (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sue Jasulaitis, RN MS Clinical Research Coordinator, Angeline Beltsos, M.D., Fertility Centers of Illinois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-019
Record Dates: First submitted 2010-05-05; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Infertility
Keywords: In-Vitro Fertilization; Donor Egg IVF
MeSH Terms: conditions — Infertility | interventions — Progesterone; Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone in Oil (Active Comparator): Donor egg recipients will begin progesterone 50 mg IM injection starting the day after donor egg fertilization, and continue daily until pregnancy results can be determined.
  If pregnant, donor egg recipient will continue progesterone 50 mg IM injections daily until approximately 9 weeks of pregnancy.
  Interventions: Drug: Progesterone in Oil
- Endometrin (Active Comparator): Donor egg recipients will begin Endometrin 100 mg per vagina three times daily starting the day after donor egg fertilization and continue until pregnancy result can be determined.
  If pregnant, donor egg recipients will continue Endometrin 100 mg TID until approximately 9 weeks of pregnancy.
  Interventions: Drug: Endometrin

INTERVENTIONS:
Drug: Endometrin — 100 mg per vagina TID
  Arms: Endometrin
Drug: Progesterone in Oil — 50 mg IM injection daily
  Arms: Progesterone in Oil

SUMMARY:
The aim of this study is to evaluate both pharmaceutical therapy and advanced treatment techniques for infertile patients requiring in-vitro fertilization utilizing donor eggs.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical pregnancy rate of micronized progesterone (Endometrin, Ferring Pharmaceuticals) compared to progesterone in oil injections in in-vitro fertilization (IVF) donor egg recipients. The secondary objective is to evaluate the effectiveness of freezing/vitrification of donor eggs. Effectiveness of vitrification will be evaluated by egg thaw/survival, fertilization, and implantation rates.

ELIGIBILITY:
Inclusion Criteria:

Oocyte Donors:

* Age 21-34 years of age
* BMI 18-34
* Normal ovarian reserve, defined as FSH <10 and AFC >10
* Medical evaluation consistent with FDA criteria for donor inclusion

Donor Oocyte Recipients

* Documented history of infertility requiring donor oocyte for optimal fertility potential
* Documentation of a normal uterine cavity by hysteroscopy, hysterosonogram, or HSG within 1 year of study screening
* Fresh or Frozen Sperm

Exclusion Criteria:

Oocyte Donors:

* Abnormal ovarian reserve, defined as FSH <10, AFC>10, prior poor response to controlled ovarian hyper-stimulation(COHS)
* Failure to meet FDA criteria for donor approval (risk factor and medical evaluation)
* Previous history of poor response to COHS

Donor Oocyte Recipients:

* Uncontrolled hypothyroidism, hyperprolactinemia, or systemic disease that may interfere with study treatment
* Active thrombophlebitis or thromboembolic disorders, or a history of hormone associated thrombophlebitis or thromboembolic disorders
* Surgically aspirated sperm (TESE)
* 2 or more clinical pregnancy losses (excluding aneuploidy for previous autologous cycles)
* Clinically significant gynecologic pathology or uterine abnormality, such as submucosal fibroids > 5 cm, communicating hydrosalpinx, uncorrected uterine septum, undiagnosed vaginal bleeding, endometrial atypia, or any other condition that could adversely affect pregnancy outcomes
* History of 2 or more failed IVF donor cycles

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate of micronized vaginal progesterone (Endometrin, Ferring Pharmaceuticals) compared to intramuscular progesterone supplementation for luteal phase support after IVF-ET from previously vitrified donor eggs | 10-12 days post IVF-ET

SECONDARY OUTCOMES:
Evaluation of the effectiveness of vitrification of IVF donor oocytes. Effectiveness will be evaluated by ooctye thaw/survival rates, fertilization and implantation rates assessed from the day of oocyte thawing through IVF cycle outcome. | six to eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angeline Beltsos, MD, Principal Investigator — Fertility Centers of Illinois
Locations (1):
- Fertility Centers of Illinois, Chicago, Illinois, United States